CLINICAL TRIAL: NCT06406634
Title: Cadonilimab in Combination With Lenvatinib and Hepatic Arterial Infusion Chemotherapy (HAIC) for the Treatment of Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-M-0035
Record Dates: First submitted 2024-04-07; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cadonilimab; Lenvatinib; Hepatic Arterial Infusion Chemotherapy (HAIC); Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Cadonilimab +Lenvatinib+Hepatic Arterial Infusion Chemotherapy (HAIC) (Experimental): HAIC(FOLFOX)+Cadonilimab (AK104) (10 mg/kg, Q3W, iv) + Lenvatinib (8 mg (if patient body weight was <60 kg) or 12 mg (if patient body weight was ≥60 kg) )
  Interventions: Drug: Cadonilimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Cadonilimab — Injectable solution
  Other Names: AK104
Drug: Lenvatinib — capsule

SUMMARY:
This study is an open-label, multicenter, single-arm Phase II clinical study to evaluate the effectiveness of Cadonilimab(AK104) in Combination With Lenvatinib and Hepatic Arterial Infusion Chemotherapy (HAIC) for the Treatment of Unresectable Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. The written informed consent form should be signed before a subject participates in the trial；
2. Histologically/cytologically confirmed HCC or cirrhosis meeting the clinical diagnostic criteria of HCC by the American Association for the Study of Liver Diseases (AASLD)；
3. According to the Chinese Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2022 edition), eligible for China liver cancer staging (CNLC) Stage IIIa and is not suitable for radical treatment, such as resection, ablation, or liver transplantation. Suitable for HAIC surgery and chemotherapy drugs prescribed in advance by the research center, without any contraindications to HAIC surgery and chemotherapy drugs；
4. Child-Pugh A or B；
5. at least 1 measurable lesion according to RECIST v1.1；
6. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1；
7. Adequate organ and marrow function, as defined below； 1) Absolute neutrophil count (ANC) ≥1.5x109/L without granulocyte colony-stimulating factor in the last 14 days； 2) Platelets ≥75×109/L without transfusion in the last 14 days； 3) Hemoglobin ≥8.5 g/dL without transfusion or erythropoietin use in the last 14 days； 4) Serum total bilirubin (TBL) ≤2 × ULN； 5) AST and ALT ≤5× ULN； 6) Serum creatinine ≤1.5 × upper limit of normal (ULN)； Urine protein ≤(++) , or 24-hour urine protein quantification less than 1 g； 7) Good coagulation, defined as the international normalized ratio (INR) ≤ 2， or activated partial prothrombin time (PT) ≤ 1.5 times ULN；
8. a woman of childbearing potential (WOCBP) who is sexually active with a nonsterilized male partner must have a negative pregnancy test at the Screening visit (within 3 days before the first dose of the investigational product [Cycle 1 Day 1]). If a negative urine pregnancy test result cannot be confirmed, a blood pregnancy test will be requested. Females not of childbearing age were defined as being at least 1 year postmenopausal or having undergone surgical sterilization or hysterectomy；
9. If there is a risk of conception, all subjects (male or female) will be required to use contraception with an annual failure rate of less than 1% for the entire treatment period up to 120 days after administration of the study drug at the end of treatment；

Exclusion Criteria:

1. Containing components such as fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma that have been previously confirmed by histology/cytology;
2. Recurrence of previous hepatocellular carcinoma；
3. Autoimmune hepatitis (requires liver puncture)
4. Have a history of hepatic encephalopathy or liver transplantation;
5. Diffuse liver cancer;
6. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage;
7. History of kidney disease or nephrotic syndrome;
8. Presence of bleeding events from esophageal or gastric varices caused by portal hypertension within the past 6 months. Presence of known severe (G3) varicose veins in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator;
9. Any arterial/venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism. Presence of implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, barring stable thrombosis following the conventional anticoagulation treatment. Prophylactic use of low-dose low-molecular-weight heparin is permitted;
10. Presence of any life-threatening bleeding events;
11. consecutive dosing of aspirin or other drugs, e.g., dipyridamole and clopidogrel, known to inhibit the platelet function before the first dose;
12. Uncontrolled hypertension (systolic greater than 140 mmHg or diastolic greater than 90 mmHg) after the optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
13. Symptomatic congestive cardiac failure (NYHA Class II-IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected Qtc > 500 ms (calculated using Fridericia formula) during screening.
14. History of gastrointestinal perforation and/or fistula, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months.
15. Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures. Receipt of tissue biopsy or other minor surgeries within 7 days before the first dose, barring venipuncture and catheterization for intravenous infusion.
16. History or current experience of pulmonary fibrosis and such lung diseases as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired lung function.
17. Acute or chronic active hepatitis B or C infection
18. Active tuberculosis (TB), currently receiving anti-tuberculosis treatment or received such therapy within 1 year before the first dose.
19. Human immunodeficiency virus (HIV) infected (HIV 1/2 antibody positive) and known syphilis infection requiring treatment.
20. Active or poorly clinically controlled serious infections. Severe infections within 4 weeks before the first dose, including but not limited to hospitalization caused by infection, bacteremia, or severe pneumonia complication.
21. Receipt of immunosuppressants within 4 weeks before the first dose;
22. Receipt of a live attenuated vaccine within 4 weeks before the first dose or planned to receive a live attenuated vaccine during the study;
23. Receipt of systemic treatment with traditional Chinese medicines with cancer indications or immunomodulators (including thymosin, interferon, and interleukin, barring local use for controlling pleural fluid or ascites) within 2 weeks before the first dose;
24. Prior exposure to any agent targeting T cell costimulation or immune checkpoint pathways (e.g., anti-PD 1, anti-PD L1, anti-PD L2, anti-CTLA 4, anti CD137 or anti-OX40 antibody, etc).
25. Known allergy or reaction to any component of the Cadonilimab formulation;
26. Receipt of treatment in other clinical trials within 4 weeks before the first dose;
27. Pregnant or breastfeeding female patients;
28. Considered ineligible for participating in the trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and PR

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Time Frame: from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD
Duration of Response(DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first
Overall Survival(OS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of death due to any cause
Adverse event (AE) | From the subject signs the ICF to 90 days after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China